CLINICAL TRIAL: NCT00532636
Title: Head Position Angles in Children to Open the Upper Airway
Brief Title: Head Position Angles in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment completed
Sponsor: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AN2439
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Airway; Airway obstruction; Mouth-to-mask resuscitation; Respiration artificial; Ventilation; Ventilation of an unprotected airway; Safety and efficiency of mask ventilation; Avoidance of stomach inflation
MeSH Terms: conditions — Airway Obstruction; Respiratory Aspiration | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Children 1-5 years of age
  Interventions: Procedure: Ventilation
- 2 (Active Comparator): Children 6-10 years of age
  Interventions: Procedure: Ventilation

INTERVENTIONS:
Procedure: Ventilation — Mask ventilation in neutral and head extension position
  Arms: 1
Procedure: Ventilation — Mask ventilation in neutral and head extension position

SUMMARY:
Inexperienced rescuers may encounter severe problems in an unconscious patient in opening and maintaining an upper airway patent. Designing a ventilating device that could indicate how to open an upper airway correctly may be beneficial. The head of children is randomly placed in different head positions by one investigator. A ventilating mask is then pressed gently on the child's face followed by measurement of the head position angles and pulmonary function. This information could be utilised to optimise assisted ventilation of an unprotected upper airway in children.

DETAILED DESCRIPTION:
Ventilation during basic life support improves survival in cardiac arrest patients significantly. Unfortunately, this is in contrast to the willingness of potential rescuers to perform mouth-to-mouth ventilation. For example, although healthcare professionals would perform mouth-to-mouth ventilation on a 4-year old drowned child in >90% of cases, this likelihood would decrease to ~10% in the case of a young male unconscious patient in a San Francisco public bus. Possibly, lay rescuers would perform assisted ventilation more often if a simple ventilation device were available. However, both the willingness to perform assisted ventilation plus the ability to open and to maintain the airway patent are necessary to ensure efficient ventilation in an unconscious patient with an unprotected upper airway.

Since retention of skills after basic life support classes are notoriously low, a resuscitation tool should incorporate self-explanatory features to improve applicability, and to provide built-in safety. Thus, an option could be to ensure an open airway by the use of a built-in indicator within a ventilating device to confirm correct head extension. One possible approach may be to determine head positions that make an open airway likely, and then extrapolate these angles to a scale that could be integrated into a ventilating device; however, safe head extension needs to be determined first to prevent harm. The purpose of this study is to determine head position angles reflecting neutral position and maximal extension in unconscious supine children in a first step to design a ventilating device to optimise ventilation of an unprotected upper airway.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II children, 1-10 years of age

Exclusion Criteria:

* Facial deformity
* Pathological airway or cervical spine
* BMI>35
* History of gastric reflux

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Wenzel, Prof., MD, MSc, Study Chair — Dept. of Anesthesia and Critical Care Medicine
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

REFERENCES:
- [Derived] Paal P, Niederklapfer T, Keller C, von Goedecke A, Luckner G, Pehboeck D, Mitterlechner T, Herff H, Riccabona U, Wenzel V. Head-position angles in children for opening the upper airway. Resuscitation. 2010 Jun;81(6):676-8. doi: 10.1016/j.resuscitation.2010.01.022. Epub 2010 Mar 26. PMID 20346568